CLINICAL TRIAL: NCT02935881
Title: A Prospective Randomized Trial Comparing Endoscopic Radio Frequency Ablation (RFA) - STRETTA vs Sham Therapy for the Treatment of Refractory Gastroesophageal Reflux Disease
Brief Title: STRETTA ,Radio Frequency Ablation (RFA) v/s Sham Therapy for the Treatment of Refractory GERD
Acronym: STRETTAGERD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Rakesh K, consultant gastroenterologist, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aigstretta 001
Record Dates: First submitted 2016-10-11; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA (Stretta Procedure) (Active Comparator): Radio Frequency Ablation (RFA) using a Stretta device.
  Interventions: Device: Radio Frequency Ablation (RFA) (Stretta Procedure)
- Placebo Arm (Sham Comparator): Stretta device used but RFA will not be generated.
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Device: Radio Frequency Ablation (RFA) (Stretta Procedure) — Radio Frequency Ablation (RFA) for the treatment of refractory gastroesophageal reflux disease.
  Arms: RFA (Stretta Procedure)
Procedure: Sham Procedure — Stretta device will be used but Radio Frequency Ablation (RFA) will not be generated.
  Arms: Placebo Arm

SUMMARY:
Gastro-esophageal reflux disease (GERD) is a chronic disorder with significant impact on the quality of life of patients. It may also lead to several complications like peptic strictures, ulcerations, Barrett 's disease and subsequently adenocarcinoma of the esophagus. Proton pump inhibitors (PPIs) are the mainstay of GERD treatment, with up to 90 % of patients with reflux disease becoming asymptomatic while taking PPIs. Several studies have demonstrated that RF delivery at the gastro-esophageal junction(GEJ), also called the Stretta procedure, induces symptom relief and decreases need of PPI intake in GERD. The investigators propose to perform a sham-controlled randomized study to evaluate the influence of the Stretta procedure on symptoms and esophageal acid exposure in patients of refractory GERD.

DETAILED DESCRIPTION:
Gastro-esophageal reflux disease (GERD) is a chronic disorder with significant impact on the quality of life of patients. It may also lead to several complications like peptic strictures, ulcerations, Barrett 's disease and subsequently adenocarcinoma of the esophagus. Proton pump inhibitors (PPIs) are the mainstay of GERD treatment, with up to 90 % of patients with reflux disease becoming asymptomatic while taking PPIs. However, the treatment of patients with proven GERD, who have an unsatisfactory response to high doses of PPIs remains a challenge. A number of endoscopic procedures, aimed at improvement of the barrier function of the lower esophageal sphincter (LES), have emerged over the last decade. Several studies have demonstrated that RF delivery at the gastro-esophageal junction(GEJ), also called the Stretta procedure, induces symptom relief and decreases need of PPI intake in GERD. The investigators propose to perform a sham-controlled randomized study to evaluate the influence of the Stretta procedure on symptoms and esophageal acid exposure in patients of refractory GERD.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18years
* Small hiatus hernia (< 2-3 cm)
* Los Angeles Grade 'A' or 'B' Reflux Esophagitis
* LES pressure : 5 - 15 mm Hg
* PPI dependent / refractory GERD
* 24 hr acid exposure study showing abnormal esophageal acid exposure > 4%
* DeMeester Score >14.7
* Esophageal manometry showing normal peristalsis

Exclusion Criteria

* Age < 18 years
* Large hiatus hernia (> 3 cm)
* Los Angeles Grade 'C' or 'D' Reflux Esophagitis
* LES pressure : < 5 or > 15 mm Hg
* Underlying coagulation disorder
* Previous Esophageal or Gastric surgery
* H/o coronary artery disease (CAD)
* Esophageal manometry showing ineffective peristalsis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients who report improvement in Quality of Life (QOL) post Stretta procedure as compared to Sham therapy. | 1 year
  6 point GERD Likert Scale will be used to assess the improvement in frequency and severity of GERD symptoms post Stretta procedure & Sham therapy amongst patients.

SECONDARY OUTCOMES:
Number of patients who report independence from Proton Pump Inhibitor (PPI) drug post Stretta procedure as compared to Sham therapy. | 1 year
  Questionnaire will be provided to each participant to report no further requirement of PPI drug post procedure.
Comparison of Increased Lower Esophageal Sphincter pressure among patients post Stretta procedure & Sham Therapy. | 1 year
  High Resolution Esophageal Manometry will be performed after the procedure in each patient to compare the LES pressure between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kalapala Rakesh, MD,DM, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian insititute of gastroenterology somajiguda, hyderabad india, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No